CLINICAL TRIAL: NCT00429949
Title: A Phase II Study of Dasatinib in the Treatment of Relapsed or Plateau Phase Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-1159
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Relapsed, Refractory or Plateau Phase Multiple Myeloma
Keywords: Dasatinib; Plateau phase
MeSH Terms: conditions — Recurrence | interventions — Dasatinib

ARMS (1):
- Dasatinib (Experimental): Dasatinib will be administered continuously at an oral dose of 70 mg BID on Days 1-28 of each 28 day cycle.
  In patients with stable disease after 8 weeks on therapy the dasatinib will be increased to 100 mg BID on Days 1-28 on each 28 day cycle.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib
  Other Names: Sprycel

SUMMARY:
To evaluate the response rate (Complete Response [CR] and Partial Response [PR]) to dasatinib in patients with relapsed, refractory or plateau phase multiple myeloma whose serum paraprotein levels are >0.5g/dL or urine paraprotein levels are >1.0g/24 hours.

DETAILED DESCRIPTION:
Studies have confirmed the ability of dasatinib to inhibit numerous kinases (76 of 148 kinases tested in one series).13 Overexpression or dysregulation of a number of kinases have been implicated in the pathophysiology of MM and could serve as potential targets for inhibition by dasatinib.

Fibroblast growth factor 3 (FGFR3), which is not normally expressed in plasma cells, is aberrantly expressed in 15 % of multiple myeloma patients. Its expression results from the translocation t4;14.14 Dasatinib weakly inhibits FGFR3.13

Another target for inhibition in multiple myeloma is the epidermal growth factor receptor family, particularly ErbB4. In vitro, ErbB4 was expressed in 4 of 9 myeloma cell lines, and a panErbB inhibitor induces apoptosis in myeloma cell lines.15 Dasatinib has been shown to have moderate affinity for ErbB4.13

Members of the src family of protein-tyrosine kinases are also potential targets for therapy in multiple myeloma. Hematopoietic cell kinase (Hck) is a src family member whose expression is restricted to hematopoietic cells of the myeloid and B-lymphoid lineages. Hck mediates IL-6 induced proliferative signals, which are potent growth and survival factors in multiple myeloma.16 Lyn and Fyn are two additional src family protein-tyrosine kinases that may serve as targets for therapy in myeloma. Lyn is strongly expressed in myeloma cell lines, while Fyn expression is variable. Activation of Lyn and Fyn appears requisite to IL-6-induced proliferation.17 Selective inhibition of Lyn in vitro suppresses IL-6 induced proliferation.18 Dasatinib has high affinity for both Fyn and Lyn, and inhibition may reduce IL-6 induced proliferation.13

The receptor tyrosine kinase c-kit is overexpressed in one-third of cases of multiple myeloma. 19 Inhibition of c-kit with imatinib results in inhibition of proliferation in vitro.20 Unfortunately, in a phase II clinical study of imatinib in relapsed/refractory myeloma, there were no responses.21 However, dasatinib binds c-kit with greater avidity than does imatinib.13

Myeloma cells are heterogeneous in their biological characteristics, such as their proliferative response to IL-6, as well as their immunophenotypes, including CD45 expression. The promiscuous nature of kinase inhibition by dasatinib may tolerate small changes in the kinase and remain able to inhibit mutant kinases.

In addition to potential antimyeloma effects of dasatinib, there are potentially additional benefits. Src plays an essential role in osteoclast function and bone resorption.22 As a Src inhibitor, dasatinib inhibits bone resorption in vitro. 11 Src inhibition by dasatinib in patients with multiple myeloma could produce beneficial effects on bone density.

We propose a single-arm, phase II, open-label study of dasatinib in patients with relapsed or plateau-phase multiple myeloma.

ELIGIBILITY:
Inclusion Criteria

* Multiple myeloma diagnosed by standard criteria with either relapsed or plateau-phase disease.

  * Relapsed: At least 1 prior therapy for multiple myeloma with documented evidence of progression on the most recent treatment.
  * Plateau-phase: subjects with myeloma who had a response to their most recent multiple myeloma therapy (including autologous transplantation or other investigational agents) and have residual detectable monoclonal protein in their serum or urine that has been stable for greater than or equal to 3 months (+/- 25% change in M-protein).
* Measurable levels of monoclonal protein in serum (greater than or equal to 0.5 g/dL) or urine (greater than or equal to 1.0 g/24 hr).
* Age 18 years or older.
* ECOG performance status of less than or equal to 2.
* Acceptable organ and marrow function as defined below:

  * Hemoglobin of greater than or equal to 8 gm/dL
  * Absolute neutrophil count of greater than or equal to 500/mm3
  * Platelets of greater than or equal to 50,000/mm3
  * PT and PTT of less than or equal to 1.5 times the institutional Upper Limit of Normal (ULN)
  * Total bilirubin of less than or equal to 2.0 times the institutional ULN institutional ULN
  * Hepatic enzymes (AST, ALT ) equal to 2.5 times the institutional ULN
  * Serum Na, K+, Mg2+, Phosphate and Ca2+ greater than or equal to Lower Limit of Normal (LLN)
  * Serum Creatinine of less than or equal to 1.5 times the institutional ULN
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to take oral medication (dasatinib must be swallowed whole)
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (sensitivity of less than or equal to 25IU HCG/L) within 72 hours prior to the start of study drug administration
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped.
* Signed written informed consent including HIPAA according to institutional guidelines.

Exclusion Criteria

* Receiving any of the following therapies or medications:

  * Any investigational agents within 30 days.
  * Drugs that are generally accepted to have a risk of causing Torsade de Pointes including:
  * quinidine, procainamide, disopyramide
  * amiodarone, sotalol, ibutilide, dofetilide
  * erythromycin, clarithromycin
  * chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone,
  * halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
  * Subjects who have discontinued any of these medications must have a wash-out period of at least 7 days prior to the first dose of dasatinib.
  * Medications known to be potent CYP3A4 inhibitors (See Appendix D).
  * The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy (See section 5.5.2.3 for important cautions regarding use of antacids.)
  * Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy.
  * Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
  * Prior therapy with dasatinib
* Biopsy proven amyloidosis.
* History of other malignancy (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) which required radiotherapy or systemic treatment within the past 5 years.
* Concurrent medical condition which may increase the risk of toxicity, including:

  * Pleural or pericardial effusion of any grade
  * Clinically-significant coagulation or platelet function disorder (e.g. known von Willebrand's disease)
* Cardiac Symptoms or Cardiovascular Disease, including:

  * Myocardial infarction within 6 months
  * Uncontrolled angina within 6 months
  * Congestive heart failure within 6 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes). Any subject with a history of any arrhythmia should be discussed with the Investigator prior to entry into the study.
  * Prolonged QTc interval on pre-entry electrocardiogram (greater than 450 msec) on Bazett's correction. However, if Bazett's correction is high (i.e., greater than 450 msec) and Fridericia is less than or equal to 450 msec, the subject is eligible.
  * Subjects with hypokalemia or hypomagnesemia if it cannot be corrected
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorder (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (less than or equal to 3 months) significant gastrointestinal bleeding
* Women:

  * are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or
  * have a positive pregnancy test at baseline, or
  * are breastfeeding.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Sexually active women of childbearing potential (WOCBP) must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.

Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.

All WOCBP MUST have a negative pregnancy test prior to first receiving dasatinib. If the pregnancy test is positive, the patient must not receive dasatinib and must not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington Universtiy
Locations (1):
- Washington Universtiy in St. Louis, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib: Dasatinib will be administered continuously at an oral dose of 70 mg BID on Days 1-28 of each 28 day cycle.
Period: Overall Study
Arm/Group | Dasatinib
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 59 [38 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 21
Durie-Salmon Stage [Number; unit: participants] — Stage I: Hemoglobin (Hb) > 10g/dL, normal calcium, normal or single plasmacytoma or osteoporosis, Serum paraprotein level < 5 g/dL if IgG, < 3 g/dL if IgA, Urinary light chain excretion < 4 g/24h Stage 2: Not fufilling criteria of Stage I or III Stage III: Hb < 8.5g/dL, calcium > 12 mg/dL, 3 or more lytic bone lesions, Serum paraprotein > 7g/dL if IgG, > 5 g/dL if IgA, Urinary light chain excretion > 12g/24h
  Stages I, II, and III can be divided into A or B depending on serum creatinine:
  A: serum creatinine < 2 mg/dL (< 177 μmol/L) B: serum creatinine > 2 mg/dL (> 177 μmol/L)
  participants
    Stage IA | 2
    Stage IIA | 3
    Stage IIIA | 15
    Stage IIIB | 1
Prior therapies [Median (Full Range); unit: therapies] | 3 [1 to 14]
Prior therapies [Number; unit: participants]
  Immunomodulatory agents | 19
  Bortezomib | 10
  Anthracycline-containing regimens | 12
  Prior autologous stem cell transplant | 19
Beta 2 microglobulin at study entry [Median (Full Range); unit: mg/L] | 2.7 [1.2 to 13]
Disease status at study entry [Number; unit: participants]
  Relapsed | 14
  Plateau phase | 7
Paraprotein [Number; unit: participants]
  IgG | 14
  IgA | 6
  Light chain only | 1
Cytogenetics [Number; unit: participants]
  Normal | 12
  Del 13/13q | 2
  Complex (including 1 with t4;14) | 2
  t9;16 | 1
  Del 6p | 1
  Unavailable | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate [Complete Response (CR) and Partial Response (PR)]
Description: CR requires all of the following:
  * Absence of the original monoclonal paraprotein in serum and urine by immunofixation, maintained for a minimum of 6 weeks. The presence of oligoclonal bands consistent with oligoclonal immune response reconstitution does not exclude CR.
  * < 5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy, if biopsy is performed. If absence of monoclonal protein is sustained for 6 weeks it is not necessary to repeat the bone marrow.
  * No increase in the size or number of lytic bone lesions (development of a compression fracture does not exclude response).
  * Disappearance of soft tissue plasmacytoma
  PR requires all of the following:
  * 50% reduction in the level of the serum monoclonal paraprotein maintained for a minimum of 6 weeks.
    -Reduction in 24 hr urinary light chain excretion by either > 90% or to < 200 mg, maintained for a minimum of 6 weeks.
  * 50% reduction in the size of soft tissue plas
Time Frame: Completion of treatment (median duration of therapy was 51 days)
Measure: Number; unit: participants
Groups:
- Dasatinib 70 mg BID: Dasatinib will be administered continuously at an oral dose of 70 mg BID on Days 1-28 of each 28 day cycle.
- Dasatinib 100 mg BID: In patients with stable disease after 8 weeks on therapy the dasatinib will be increased to 100 mg BID on Days 1-28 on each 28 day cycle.
Arm/Group | Dasatinib 70 mg BID | Dasatinib 100 mg BID
Number analyzed (Participants) | 21 | 6
participants
  Complete response | 0 [0.5 to 17.3] | 0
  Partial response | 0 | 1

2. Secondary Outcome: Time to Response
Description: Time to response is measured from the start of treatment until the first date that criteria are met for complete response or partial response.
Time Frame: Completion of treatment (median duration of therapy was 51 days)
Population: Only one patient achieved a partial response.
Measure: Number; unit: cycles
Arm/Group | Dasatinib
Number analyzed (Participants) | 1
cycles | 5

3. Secondary Outcome: Safety and Tolerability of Dasatinib (Grade III-IV Toxicities)
Description: Toxicities were graded using the NCI Common Toxicity Criteria v3.0.
Time Frame: Up to 30 days following end of treatment (median duration of therapy was 51 days)
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 21
participants
  Grade III anemia | 5
  Grade III neutropenia | 2
  Grade III thrombocytopenia | 2
  Grade IV thrombocytopenia | 3
  Grade III epistaxis | 2
  Grade III gastrointestinal bleed | 1
  Grade III acute renal failure | 2
  Grade III headache | 1
  Grade III aphasia due to laryngeal plasmacytoma | 1
  Grade III neuropathy | 1
  Grade III fatigue | 1
  Grade III hypertension | 1
  Grade III diarrhea | 1
  Grade III leg/hip pain | 1
  Grade III generalized pain | 3
  Grade III hypercalcemia | 1
  Grade IV hypoglycemia | 1
  Grade IV hyperglycemia | 1
  Grade III pneumonia | 3
  Grade III pulmonary edema | 1
  Grade III pneumonitis/pulmonary infiltrates | 2
  Grade III pulmonary hypertension | 1
  Grade III hypoxia | 1
  Grade III dyspnea | 1
  Grade IV dyspnea | 1

4. Secondary Outcome: Duration of Response
Description: Duration of response is measured from the first date that criteria are met for complete response or partial response until the first date that criteria for relapse or progressive disease are met.
Time Frame: Completion of treatment (median duration of therapy was 51 days)
Population: Only one patient achieved a partial response.
Measure: Number; unit: cycles
Arm/Group | Dasatinib
Number analyzed (Participants) | 1
cycles | 3

5. Secondary Outcome: Event-free Survival (EFS) for Participants With Plateau Phase Disease
Description: EFS is defined as time from the start of the treatment until the first date that criteria for progressive disease are met, therapy was discontinued for toxicity, or death, whichever occurs first. Those patients alive will be censored at the date of last clinical contact. If progression is based upon serum or urine paraprotein measurements, which must be repeated for confirmation, event-free progression is still measured from the start of treatment until the first date that progression is detected.
Time Frame: Completion of treatment (median duration of therapy was 51 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dasatinib
Number analyzed (Participants) | 7
days | 138 [73.8 to 202.2]

6. Secondary Outcome: Event-free Survival (EFS) for Participants With Relapsed Disease
Description: as for outcome 5
Time Frame: Completion of treatment (median duration of therapy was 51 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dasatinib
Number analyzed (Participants) | 14
days | 31 [23.7 to 38.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment until 30 days following the completion of treatment (median duration of therapy was 51 days)
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=21)
Death due to disease progression (General disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Febrile neutropenia (Infections and infestations) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathy - motor (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=21)
Alkaline phosphatase (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Aphasia (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Ataxia (Nervous system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bad dreams (Psychiatric disorders) | 1
Bone ache (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Buttocks pain (Musculoskeletal and connective tissue disorders) | 1
Catheter-related infection (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Decubitus ulcer - sacral (Skin and subcutaneous tissue disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Diaphoresis (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Distension (Gastrointestinal disorders) | 4
Dizziness/lightheadedness (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 2
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Ears "clogged" (Ear and labyrinth disorders) | 1
Ears "popping" (Ear and labyrinth disorders) | 1
Edema - limbs (General disorders) | 7
Elevated creatinine (Investigations) | 3
External ear pain (Ear and labyrinth disorders) | 1
Eye bleed (Eye disorders) | 1
Face/brow pain (Musculoskeletal and connective tissue disorders) | 1
Facial bumps (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 12
Fever (General disorders) | 8
Flatulence (Gastrointestinal disorders) | 1
Foot pain (Musculoskeletal and connective tissue disorders) | 1
Gastric irritation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Generalized pain (General disorders) | 4
Gritty sensation in mouth (Gastrointestinal disorders) | 1
Gynecomastia (Endocrine disorders) | 1
Head pressure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Heel pain (Musculoskeletal and connective tissue disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 11
Hip pain (Musculoskeletal and connective tissue disorders) | 2
Hot flashes (Vascular disorders) | 3
Hypercalcemia (Investigations) | 2
Hyperglycemia (Investigations) | 3
Hypermagnesemia (Investigations) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypertension (Cardiac disorders) | 2
Hypervolemia (Blood and lymphatic system disorders) | 3
Hypoalbuminemia (Investigations) | 4
Hypocalcemia (Investigations) | 2
Hypoglycemia (Investigations) | 3
Hypokalemia (Investigations) | 1
Hypomagnesemia (Investigations) | 1
Hyponatremia (Investigations) | 5
Hypotension (Cardiac disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Incontinence (Renal and urinary disorders) | 2
Infection without neutropenia (Infections and infestations) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 2
Leukocytes (Investigations) | 5
Lower GI bleed (Gastrointestinal disorders) | 1
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 3
Lymphocele (cyst on face) (Blood and lymphatic system disorders) | 1
Lymphopenia (Investigations) | 11
Mood alteration - anxiety (Psychiatric disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Neuropathy - motor (Nervous system disorders) | 3
Neuropathy - sensory (Nervous system disorders) | 3
Neutrophils (Investigations) | 4
Night sweats (General disorders) | 2
Nipple pain (Musculoskeletal and connective tissue disorders) | 1
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 2
Odor (patient odor) (General disorders) | 1
Oily face (Skin and subcutaneous tissue disorders) | 1
Oral/gum/teeth pain (Gastrointestinal disorders) | 2
Petechiae (Blood and lymphatic system disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelets (Investigations) | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Renal failure (Renal and urinary disorders) | 2
Right side of nose swollen (General disorders) | 1
Rigors (General disorders) | 3
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1
SGOT (AST) (Investigations) | 5
SGPT (ALT) (Investigations) | 3
Sensitive teeth (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Sinus discharge (Respiratory, thoracic and mediastinal disorders) | 1
Sinus infection (Infections and infestations) | 1
Skin tears (Injury, poisoning and procedural complications) | 1
Somnolence (Nervous system disorders) | 1
Stomach tightness (Gastrointestinal disorders) | 1
Tachycardia (Cardiac disorders) | 2
Thigh pain (Musculoskeletal and connective tissue disorders) | 1
Tongue felt "thick" (Gastrointestinal disorders) | 1
Under tongue felt swollen (Gastrointestinal disorders) | 1
Upper extremity pain (Musculoskeletal and connective tissue disorders) | 2
Upper respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 2
Uric acid (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes